CLINICAL TRIAL: NCT03135535
Title: Micro-mobile Foot Compression Device to Improve Motor-function in People With Diabetes and Loss of Protective Sensation
Brief Title: Micro-mobile Foot Compression and Diabetic Foot
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Avex LLC (Industry)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Professor of Surgery, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H-37962
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Results first posted 2020-02-27 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Diabetes; PAD; Lower Extremity Edema; Neuropathy;Peripheral; Foot Ulcer, Diabetic; Lymphatic Diseases
MeSH Terms: conditions — Diabetes Mellitus; Neuritis; Diabetic Foot; Lymphatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Avex Footbeat (Experimental): Subjects will receive a new pair of diabetic shoes with BOA shoelace closure and a pair of AVEX Footbeat insoles, which include a micro-mobile compression pump. The entire system is named 'intervention shoes' for simplicity. They will be instructed to wear the intervention shoes on daily basis for 4 weeks for duration of at least 4 hours per day.
  Interventions: Device: Avex Footbeat

INTERVENTIONS:
Device: Avex Footbeat — Subjects will receive diabetic shoes equipped with Boa Technology shoelace system and Footbeat compression insoles, which for simplicity will be named intervention shoes. All participants will be asked to wear the intervention shoes for duration of 4-weeks on daily basis (minimum 4 hours per day). Daily use of the intervention shoes will be assumed to improve balance, mobility, plantar sensation, lower extremity edema, and lower extremity skin perfusion.

SUMMARY:
Diabetic foot ulceration (DFU) is a common and largely preventable complication. While most of these ulcers can be treated successfully, some will persist and become infected. Ultimately, nearly one fifth of patients with infected lower-extremity diabetic ulcers will require amputation of the affected limb.Prevention by identifying people at higher risk is the key for better clinical management of such patients. It is not uncommon for patients suffering from diabetes to have concomitant lower extremity edema or even venous insufficiency and they subsequently may benefit from graduated compression. However, because of the common association of peripheral arterial disease (PAD) in patients with diabetes, most clinicians are reluctant to apply compressive dressings in fear of exacerbating the symptoms of PAD and the possible resulting gangrene.

A novel micro-mobile foot compression device named Footbeat (AVEX, Inc.) offers alternative means providing lower extremity compression. This device is portable and can be used in a standard diabetic shoes on daily basis, which in turn may improve venous blood and relief from concomitant lower extremity edema. In addition, potential improvement in lower extremity blood flow in response to regular foot compression, could improve balance, gait, skin perfusion, plantar sensation, and overall daily physical activities (e.g. number of taken steps per day, duration of standing, etc).

The purpose of this study is to conduct an observational study with N=30 ambulatory patients with diabetes and loss of protective sensation to assess whether this micro-mobile foot compression device can help improving motor function, lower extremity perfusion, and vascular health.

ELIGIBILITY:
Inclusion Criteria:

* Male or female , age 18 or older with the ability and willingness to provide Informed consent
* Patient is willing to participate in all procedures and follow up evaluations necessary to complete the study
* History of type 2 diabetes confirmed by patient's physician.
* History of peripheral neurpathy .

Exclusion Criteria:

* Patients with severe peripheral vascular disease (ankle-brachial systolic pressure index (ABI) <0.5 or ABI>1.30)
* Patients with active wound infection, or untreated osteomyelitis
* Patients with major foot deformities (e.g. Charcot Foot) or major amputation (e.g. above ankle)
* Unamulatory of those who are unable to independently walk with or without walking assistance, a distance of 40 feet.
* Patients who are unable or unwilling to participate in all procedures and follow up evaluations
* Patients currently on immunosuppressive drugs.
* Pregnant or breast feeding ladies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-09-09 (Actual); Study Completion 2021-05-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Only de-identified data and associated results will be published in peer-review papers or scientific abstracts. The de-identified data from changes in primary and secondary outcomes (e.g. changes in balance, gait, physical activity, edema, etc) may be shared upon approval of the sponsor.

REFERENCES:
- [Result] Kang GE, Zahiri M, Lepow B, Saleem N, Najafi B. The Effect of Daily Use of Plantar Mechanical Stimulation Through Micro-Mobile Foot Compression Device Installed in Shoe Insoles on Vibration Perception, Gait, and Balance in People With Diabetic Peripheral Neuropathy. J Diabetes Sci Technol. 2019 Sep;13(5):847-856. doi: 10.1177/1932296819839703. Epub 2019 Apr 3. PMID 30943782

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Avex Footbeat
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Avex Footbeat
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 5
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Balance From Baseline to 4 Weeks
Description: Balance will be quantified by measuring body sway in medial-lateral direction using a validated wearable sensors technology (Balansens, Biosensics LLC) and body sway change after 4-weeks of daily use of AVEX Footbeat will be assessed compare to baseline. Th unit of measurement is cm.
Time Frame: baseline and 4 weeks.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Avex Footbeat
Number analyzed (Participants) | 30
cm
  At Baseline | 0.94 (0.43)
  At 4-week | 0.76 (0.32)

2. Primary Outcome: Change in Skin Perfusion From Baseline to 4 Weeks
Description: Skin perfusion was quantified using Skin Perfusion Pressure Test (SPP) at the lower extremities at baseline and at 4-week (end point). The measurement of SPP was done using a device called Sensilase PAD-IQ (VASAMED). The unit of measurement is mmHg.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Avex Footbeat
Number analyzed (Participants) | 30
mmHg
  At Baseline | 75.1 (15.8)
  At 4-week | 75.7 (11.1)

3. Secondary Outcome: Change in Lower Extremity Edema From Baseline to 4 Weeks
Description: Edema will be measured by traditional circumference change of ankle. The unit of measurement is cm.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Avex Footbeat
Number analyzed (Participants) | 30
cm
  Baseline | 23.1 (2.6)
  @4week | 23.0 (2.4)

4. Secondary Outcome: Change in Plantar Sensation From Baseline to 4-week
Description: The change in plantar sensation after 4-weeks use of AVEX Footbeat will be assessed using vibratory perception threshold (VPT) test. The unit of this measurement is volt.
Time Frame: Baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: volts
Arm/Group | Avex Footbeat
Number analyzed (Participants) | 30
volts
  At Baseline | 27.4 (12.6)
  At 4-week | 23.3 (11.9)

5. Secondary Outcome: Change in Stride Velocity From Baseline to 4-week
Description: The change in stride velocity was quantified by gait speed measured using a validated wearable sensor (LEGSys, Biosensics, LLC). The unit of measurement is meter per second (m/s)
Time Frame: Baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Avex Footbeat
Number analyzed (Participants) | 30
m/s
  At Baseline | 0.87 (0.21)
  At 4-week | 0.96 (0.23)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Serious adverse event (SAE) was defined as any related incident of foot ulcer caused by the proposed footwear/insole
  Other adverse event (AE) was defined as any related major pain or any other problems associated with provided footwear (e.g. edema, skin redness, callus, etc)
Arm/Group | Avex Footbeat
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT03135535/Prot_SAP_001.pdf